CLINICAL TRIAL: NCT05291117
Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Apnoeic Ventilation During Operative Hysteroscopic Procedures Under General Anesthesia: an Observational Study.
Brief Title: THRIVE Ventilation for Operative Hysteroscopy Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4631
Record Dates: First submitted 2022-01-19; First posted 2022-03-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Oxygen; General Anesthesia; Hysteroscopy
Keywords: Transnasal humified high flow oxygen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) allows to extend the apnoeic window in patients undergoing general anesthesia by delivering 100% of heated and humidified oxygen at 70L/min in order to maintain viable gas exchange during an extended period of cessation of spontaneous ventilation.

This technique has been successfully applied in several clinical settings (induction of general anesthesia, laryngoscopy in predicted difficult airway management, and as unique airway management technique for procedural sedation or general anesthesia for brief surgical procedures).

Operative hysteroscopy is a brief surgical procedure usually performed under general anesthesia with intravenous agents (propofol plus fentanyl) and positive pressure ventilation through facial or laryngeal mask.

The aim of this study is to investigate the effects of THRIVE apnoeic ventilation during hysteroscopy under general anesthesia. Our primary outcome is to describe the trend of SpO2 and tcCO2 during the procedures.

Secondary outcomes include description of arrhythmias requiring medical treatment, hemodynamic instability, unmanageable copious secretions, airway obstruction or inability to maintain airway patency, witnessed aspiration, airway related complications, number of airway manipulations, adverse events, assessment of postoperative dyspnoea and comfort, patient satisfaction.

Women (> 18 years old and < 70 years old), ASA physical status I and II presenting for elective operative hysteroscopies will be included.

A number of 30 patients was planned to target the primary outcome.

DETAILED DESCRIPTION:
Background Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE), term coined by Patel and Nouraei, refers to a technique that allows to extend the apnoeic window in patients undergoing general anesthesia by delivering 100% of heated and humidified oxygen at 70L/min using the Optiflow THRIVE-TM system (Fisher and Paykel Healthcare Ltd, Auckland, New Zealand), in order to maintain viable gas exchange during an extended period of cessation of muscular activity.

Apnoeic oxygenation is a physiological phenomenon in which oxygen flow into the lungs is driven by a negative pressure gradient generated by the difference between the alveolar rates of oxygen absorption and carbon dioxide excretion.

Potentially rapid and dangerous rise in carbon dioxide concentration is prevented by the underlying mechanisms occurring during high-flow nasal oxygenation under apnoeic conditions.

As proposed by Slutsky and more recently by Hermez, cardiogenic oscillations (changes in airway gas flow and pressure synchronous with the cardiac cycle) and their interactions with supraglottic turbulence generated by high-flow nasal oxygenation might be the underlying mechanisms of THRIVE and of the enhanced clearance of carbon dioxide.

Many clinically relevant benefits have been associated with nasal high flow. It provides a constant FiO2 by delivering the gas at flow rates that exceed the patient's peak inspiratory flow rate. It is effective in providing a flow-dependent effect of continuous positive airway pressure of about 1 cmH20 for every 10 L/min increase in gas flow within a range of 30-50 L/min, up to 11.9 cm H20 at a maximum flow of 100 L/min. Moreover, it reduces respiratory rate, it clears in a dose-dependent manner dead space of the upper airways and possibly even below the soft palate, leading to a reduction in rebreathing of expired air, with the potential to increase the alveolar volume and to improve alveolar ventilation and gas exchange. It is likely that, especially in patients with mild to moderate respiratory failure, enhanced comfort from heated humidification and flushing of dead space, lessen the work of breathing, thus improving thoraco-abdominal synchrony. By contrast, in spontaneously breathing patients, as a consequence of the large amount of air inflated into the stomach, higher number of reflux events could be detected increasing the risks of aspiration.

This technique has been successfully applied in several clinical settings to extend the apnoeic window after the induction of general anesthesia and during laryngoscopy in predicted difficult airway management. As long as airway patency was present, it succeeded in extending the apnoeic window up to 65 minutes. PaO2 and peripheral oxygen saturation remained stable and the rate of rise of CO2 during apnoea was reduced from earlier findings of 0.5 kPa/min with conventional low-flow systems to 0.15 kPa/min.

THRIVE has also been used as unique airway management technique for procedural sedation or when general anesthesia was performed for brief surgical procedures: it was able to keep patients with mild systemic disease well oxygenated, maintaining PaO2 stable with decreased rates of rise of CO2 during apnoea, as compared to conventional low-flow systems for oxygen therapy, such as the Venturi mask.

Operative hysteroscopy is a brief surgical procedure (< 30 minutes), usually performed in a day-surgery regimen. Typical anesthesiologic management in this setting includes general anesthesia with intravenous agents (propofol plus fentanyl) and positive pressure ventilation through laryngeal mask (I-gel). The application of THRIVE in this setting has potential advantages either for the patient, including minimal airway manipulation and greater comfort, either for the anesthesia provider, facilitating procedural technique and airway management.

Aim of the study The aim of this study is to investigate the effects of THRIVE apnoeic ventilation during operative hysteroscopy under general anesthesia.

Monitoring Standard perioperative monitoring will include non-invasive blood pressure (NIBP) with an upper arm cuff, 3-lead ECG, peripheral oxygen saturation (SpO2) and bispectral index (BIS). NIBP will be measured every 5 minutes before induction of anesthesia and throughout the procedure. Transcutaneous carbon dioxide (tcCO2) will be continuously monitored by Radiometer TCM5 monitor.

Study protocol Upon arrival on the operating theatre, each patient will be placed in supine position in lithotomic position; a peripheral venous cannula will be inserted on the hand or forearm and 500 ml Ringer-Lactate solution infusion will be started. Omeprazole 40 mg and dexametasone 4 mg will be given preoperatively. 3 minutes of pre-oxygenation will be performed with 100% oxygen 30 L/min delivered via dedicated Optiflow THRIVE-TM nasal cannulae. General anesthesia will then be induced with target-controlled infusion (TCI) of propofol (7 mcg/kg) through Orchestra Infusion system (Fresenius Kabi) plus fentanyl (1,5 mcg/kg). The range of maintenance of propofol concentration will be 4-6 mcg/ml, titrated to maintain a level of anesthesia monitored by BIS between 40 and 50. With the onset of general anesthesia oxygen flow will be increased to 70 L/min and maintained throughout the procedure. Head repositioning, jaw thrust, oropharyngeal cannula placement could be used to improve airway patency during the procedure. In case of episodes of oxygen desaturation, defined as SpO2<94%, or rise of tcCO2 over 45 mmHg, positive pressure ventilation by facial mask or laryngeal mask will be applied by the practitioner based on clinical judgement.

At the end of the procedure, propofol will be stopped. Paracetamol 1g, ondansetron 4 mg and ketorolac 30 mg will be administered as routine clinical practice.

The awake patient will be moved to the PACU for three hours of post-operative monitoring as required by internal practice for day-surgery procedures. Standard monitoring will include NIBP measured every 15 minutes, 3-lead ECG, and peripheral oxygen saturation (SpO2).

One hour after the end of the procedure and before discharge from the PACU the patient will be asked to rate its perceived degree of dyspnoea with the Borg dyspnoea score and its degree of comfort by Visual Numerical Scale (VAS).

In case of episodes of oxygen desaturation, defined as SpO2<94%, supplemental oxygen will be initially provided to the patient by low-flow Venturi mask with FiO2 40%.

Discharge from the PACU will require an Aldrete score of 9-10.

Sample size calculation For this pilot study no sample size calculation was performed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.

Exclusion Criteria:

* BMI > 30,
* pregnancy,
* cardiac arrhythmia,
* high risk of aspiration,
* neuromuscular disease,
* patient refusal.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing operative hysteroscopy
Study Population: Women scheduled for elective operative hysteroscopies will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change of tCO2 during THRIVE ventilation. | pre-anesthesia; up to 1 hour.
  CO2 values (reported as mmHg) measured by Radiometer monitor.
change of SpO2 during THRIVE ventilation. | pre-anesthesia; up to 1 hour.
  SpO2 values (reported as "%") measured by oxymeter.

SECONDARY OUTCOMES:
Airway related complications. | 2 hours after the end of anesthesia.
  Incidence of patients requiring airway manipulations (nasal cannula, manual ventilation, laryngeal mask ventilation, tracheal intubation) by the anesthesiologist, reported as "% of total number of patients".
Postoperative complications - 1 | 2 hours after the end of anesthesia.
  Incidence of patients suffering from cough, sore throat, dysphagia, dysphonia, laryngospasm, oxygen desaturation (defined as SpO2<94%), reported as "% of total number of patients"
Postoperative complications - 2 | 2 hours after the end of anesthesia.
  Incidence of dyspnoea (measured with Borg dyspnoea score: 0= no dyspnoea, 10= maximal dyspnoea).
Postoperative complications - 3 | 2 hours after the end of anesthesia.
  Incidence of discomfort (measured with Visual Analogue Scale: 0= no discomfort, 10= maximal discomfort).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Agostino Gemelli, Rome, Italy

REFERENCES:
- [Result] BARTLETT RG Jr, BRUBACH HF, SPECHT H. Demonstration of aventilatory mass flow during ventilation and apnea in man. J Appl Physiol. 1959 Jan;14(1):97-101. doi: 10.1152/jappl.1959.14.1.97. No abstract available. PMID 13630833
- [Result] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Result] O'Cain CF, Dowling NB, Slutsky AS, Hensley MJ, Strohl KP, McFadden ER Jr, Ingram RH Jr. Airway effects of respiratory heat loss in normal subjects. J Appl Physiol Respir Environ Exerc Physiol. 1980 Nov;49(5):875-80. doi: 10.1152/jappl.1980.49.5.875. PMID 7429910
- [Result] Slutsky AS, Brown R. Cardiogenic oscillations: a potential mechanism enhancing oxygenation during apneic respiration. Med Hypotheses. 1982 Apr;8(4):393-400. doi: 10.1016/0306-9877(82)90032-9. PMID 6808323
- [Result] Hermez LA, Spence CJ, Payton MJ, Nouraei SAR, Patel A, Barnes TH. A physiological study to determine the mechanism of carbon dioxide clearance during apnoea when using transnasal humidified rapid insufflation ventilatory exchange (THRIVE). Anaesthesia. 2019 Apr;74(4):441-449. doi: 10.1111/anae.14541. Epub 2019 Feb 15. PMID 30767199
- [Result] Hernandez G, Roca O, Colinas L. High-flow nasal cannula support therapy: new insights and improving performance. Crit Care. 2017 Mar 21;21(1):62. doi: 10.1186/s13054-017-1640-2. PMID 28320436
- [Result] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Result] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405
- [Result] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Result] Chikata Y, Onodera M, Oto J, Nishimura M. FIO2 in an Adult Model Simulating High-Flow Nasal Cannula Therapy. Respir Care. 2017 Feb;62(2):193-198. doi: 10.4187/respcare.04963. Epub 2016 Nov 22. PMID 27879385
- [Result] Moller W, Feng S, Domanski U, Franke KJ, Celik G, Bartenstein P, Becker S, Meyer G, Schmid O, Eickelberg O, Tatkov S, Nilius G. Nasal high flow reduces dead space. J Appl Physiol (1985). 2017 Jan 1;122(1):191-197. doi: 10.1152/japplphysiol.00584.2016. Epub 2016 Nov 17. PMID 27856714
- [Result] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407
- [Result] Wong DT, Dallaire A, Singh KP, Madhusudan P, Jackson T, Singh M, Wong J, Chung F. High-Flow Nasal Oxygen Improves Safe Apnea Time in Morbidly Obese Patients Undergoing General Anesthesia: A Randomized Controlled Trial. Anesth Analg. 2019 Oct;129(4):1130-1136. doi: 10.1213/ANE.0000000000003966. PMID 31584919
- [Result] Mazzeffi MA, Petrick KM, Magder L, Greenwald BD, Darwin P, Goldberg EM, Bigeleisen P, Chow JH, Anders M, Boyd CM, Kaplowitz JS, Sun K, Terrin M, Rock P. High-Flow Nasal Cannula Oxygen in Patients Having Anesthesia for Advanced Esophagogastroduodenoscopy: HIFLOW-ENDO, a Randomized Clinical Trial. Anesth Analg. 2021 Mar 1;132(3):743-751. doi: 10.1213/ANE.0000000000004837. PMID 32398433
- [Result] Shih CC, Liang PC, Chuang YH, Huang YJ, Lin PJ, Wu CY. Effects of high-flow nasal oxygen during prolonged deep sedation on postprocedural atelectasis: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):1025-1031. doi: 10.1097/EJA.0000000000001324. PMID 32890016
- [Result] Itagaki T, Okuda N, Tsunano Y, Kohata H, Nakataki E, Onodera M, Imanaka H, Nishimura M. Effect of high-flow nasal cannula on thoraco-abdominal synchrony in adult critically ill patients. Respir Care. 2014 Jan;59(1):70-4. doi: 10.4187/respcare.02480. Epub 2013 Jun 4. PMID 23737548
- [Result] Kagan I, Hellerman-Itzhaki M, Neuman I, Glass YD, Singer P. Reflux events detected by multichannel bioimpedance smart feeding tube during high flow nasal cannula oxygen therapy and enteral feeding: First case report. J Crit Care. 2020 Dec;60:226-229. doi: 10.1016/j.jcrc.2020.08.005. Epub 2020 Aug 22. PMID 32882605
- [Result] Coudroy R, Frat JP, Ehrmann S, Pene F, Terzi N, Decavele M, Prat G, Garret C, Contou D, Bourenne J, Gacouin A, Girault C, Dellamonica J, Malacrino D, Labro G, Quenot JP, Herbland A, Jochmans S, Devaquet J, Benzekri D, Vivier E, Nseir S, Colin G, Thevenin D, Grasselli G, Assefi M, Guerin C, Bougon D, Lherm T, Kouatchet A, Ragot S, Thille AW; REVA Network. High-flow nasal oxygen therapy alone or with non-invasive ventilation in immunocompromised patients admitted to ICU for acute hypoxemic respiratory failure: the randomised multicentre controlled FLORALI-IM protocol. BMJ Open. 2019 Aug 10;9(8):e029798. doi: 10.1136/bmjopen-2019-029798. PMID 31401603
- [Result] Mauri T, Galazzi A, Binda F, Masciopinto L, Corcione N, Carlesso E, Lazzeri M, Spinelli E, Tubiolo D, Volta CA, Adamini I, Pesenti A, Grasselli G. Impact of flow and temperature on patient comfort during respiratory support by high-flow nasal cannula. Crit Care. 2018 May 9;22(1):120. doi: 10.1186/s13054-018-2039-4. PMID 29743098